CLINICAL TRIAL: NCT01072435
Title: Target-controlled Infusion vs Patient-controlled Sedation With Propofol in ERCP. A Randomized Prospective Clinical Trial
Brief Title: Target-controlled Infusion Versus Patient-controlled Sedation With Propofol in Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maxim Mazanikov, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: a005c; 2009-015564-34 (EudraCT Number)
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Sedation
Keywords: ERCP; patient-controlled sedation; target-controlled infusion; propofol; Sedation with propofol for ERCP; Endoscopic Retrograde Cholangiopancreatography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient-controlled sedation (Active Comparator): PCS
  Interventions: Device: Patient-controlled sedation
- target-controlled infusion (Active Comparator): TCI
  Interventions: Device: Target-controlled infusion

INTERVENTIONS:
Device: Patient-controlled sedation — Administration of short-acting anesthetic propofol via self-administration device.Single bolus-dose 1ml(10mg)of propofol,lockout time 0sec.,no background infusion or dose-limit.
  Other Names: Arcomed/Syramed AG infusion pump designed for self administration of medicines
  Arms: patient-controlled sedation
Device: Target-controlled infusion — Anaesthesiologist´s managed target-controlled infusion of short-acting anesthetic propofol
  Other Names: Arcomed/Syramed AG target-controlled infusion device.
  Arms: target-controlled infusion

SUMMARY:
Propofol is a drug of choice for deep sedation in endoscopy. Propofol can be administered in many ways: by infusion or intravenous boluses and with self-administration device (patient-controlled sedation; PCS). It is not clear which method of propofol administration would be preferable. The main objective of the trial is to compare 2 different methods of propofol administration during ERCP: patient-controlled administration(PCS) and target-controlled infusion (TCI).

DETAILED DESCRIPTION:
80 patients of age 18-75 undergoing elective ERCP will be included to the randomized non-commercial clinical trial. Exclusion criteria are: allergy to the opioids or propofol, dementia, mental retardation, severe liver or kidney insufficiency, significant heart failure or lung disease, drug addiction. The endpoints are: ease of procedures performance, complications, degree of sedation, recovery time, propofol and opioid consumption. During the procedure patients observed and treated by the anaesthesiologist and anaesthesia nurse .

ELIGIBILITY:
Inclusion Criteria:

* elective ERCP patients

Exclusion Criteria:

* allergy to propofol or opioid;
* inability to cooperate;
* ASA(American Society of Anaesthesiology)class greater than 3

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
sedation degrees | One day
patient's and endoscopist´s satisfaction, | One day
propofol consumption | One day
vital signs:oxygen saturation,blood pressure,heart rate,breathing rate | One day

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Mazanikov, MD, Principal Investigator — Helsiki University Central Hospital,Department of Anaesthesiology; Marianne Udd, MD.,PhD, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Leena Kylänpää, Docent, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Outi Lindström, MD, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Jorma Halttunen, Docent, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Martti Färkilä, Professor, Principal Investigator — Helsinki University Central Hospital,Department of Gastroenterology; Reino Pöyhiä, Docent, Study Chair — Helsinki University Central Hospital,Department of Anaesthesiology; Harri Mustonen, PhD, Principal Investigator — Department of Gastrointestinal and General Surgery, Helsinki University Central Hospital,Helsinki,Finland
Locations (1):
- Helsiki University central Hospital,Meilahti Hospital,Endoscopy unit, Helsinki, Uusimaa, Finland